CLINICAL TRIAL: NCT02751320
Title: Clinical Efficacy of Three Experimental Toothpastes Using an in Situ Caries Model
Brief Title: Efficacy of Three Toothpastes Using an in Situ Caries Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 202301
Record Dates: First submitted 2016-04-21; First posted 2016-04-26 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-07

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Sodium Citrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Experimental Dentifrice1 (Experimental): Participants will brush their natural teeth with a pre-wetted toothbrush and their assigned dentifrice for one timed minute, ensuring the enamel specimens retained within their mouths are not directly brushed. Participants should then rinse their mouths with 15ml of tap water for approximately 10s.
  Interventions: Drug: 0.425 % w/w phytate,1150ppm F
- Experimental Dentifrice 2 (Experimental): Participants will brush their natural teeth with a pre-wetted toothbrush and their assigned dentifrice for one timed minute, ensuring the enamel specimens retained within their mouths are not directly brushed. Participants should then rinse their mouths with 15ml of tap water for approximately 10s.
  Interventions: Drug: 0.85 % w/w phytate,1150ppm F
- Experimental Dentifrice 3 (Experimental): Participants will brush their natural teeth with a pre-wetted toothbrush and their assigned dentifrice for one timed minute, ensuring the enamel specimens retained within their mouths are not directly brushed. Participants should then rinse their mouths with 15ml of tap water for approximately 10s.
  Interventions: Drug: 0.85 % w/w phytate,0.3%ZnCl2 0.5% sodium citrate, 1150ppm F
- Reference Product 1 (Placebo Comparator): Participants will brush their natural teeth with a pre-wetted toothbrush and their assigned dentifrice for one timed minute, ensuring the enamel specimens retained within their mouths are not directly brushed. Participants should then rinse their mouths with 15ml of tap water for approximately 10s.
  Interventions: Other: 0 ppm F
- Reference Product 2 (Active Comparator): Participants will brush their natural teeth with a pre-wetted toothbrush and their assigned dentifrice for one timed minute, ensuring the enamel specimens retained within their mouths are not directly brushed. Participants should then rinse their mouths with 15ml of tap water for approximately 10s.
  Interventions: Drug: 1150ppm F
- Reference Product 3 (Active Comparator): Participants will brush their natural teeth with a pre-wetted toothbrush and their assigned dentifrice for one timed minute, ensuring the enamel specimens retained within their mouths are not directly brushed. Participants should then rinse their mouths with 15ml of tap water for approximately 10s.
  Interventions: Drug: 0.3%ZnCl2, 0.5% sodium citrate, 1150ppm F

INTERVENTIONS:
Drug: 0.425 % w/w phytate,1150ppm F — Participants were assigned with 1.5±0.1g twice daily dentifrice for one timed minute.
  Arms: Experimental Dentifrice1
Drug: 0.85 % w/w phytate,1150ppm F — Participants were assigned with 1.5±0.1g twice daily dentifrice for one timed minute.
  Arms: Experimental Dentifrice 2
Drug: 0.85 % w/w phytate,0.3%ZnCl2 0.5% sodium citrate, 1150ppm F — Participants were assigned with 1.5±0.1g twice daily dentifrice for one timed minute.
  Arms: Experimental Dentifrice 3
Other: 0 ppm F — Participants were assigned with 1.5±0.1g twice daily dentifrice for one timed minute.
  Arms: Reference Product 1
Drug: 1150ppm F — Participants were assigned with 1.5±0.1g twice daily dentifrice for one timed minute.
  Arms: Reference Product 2
Drug: 0.3%ZnCl2, 0.5% sodium citrate, 1150ppm F — Participants were assigned with 1.5±0.1g twice daily dentifrice for one timed minute.
  Arms: Reference Product 3

SUMMARY:
This will be a single-centre, randomized, blinded, placebo-controlled, 6-treatment, 4-period crossover, incomplete block design, in situ caries study in healthy adults who wear a removable bilateral mandibular partial denture. The denture will be modified to accommodate 4 gauze-covered specimens of human dental enamel (4x3mm) that have been previously demineralized in vitro to form either S or low-R lesions (2 specimens of each lesion type will be used with each participant). After 14 days of twice daily product use off-site, the 2 S lesion specimens will be removed at the study site, with the remaining 2 low-R lesion specimens removed at the study site after a further 14 days of product use. To determine the remineralization ability of the treatments, all specimens will be analyzed by transverse microradiography (TMR) and enamel fluoride uptake (EFU), with the S lesions additionally analyzed by surface micro hardness (SMH) and the low-R lesions additionally analyzed by quantitative light fluorescence (QLF).

ELIGIBILITY:
Inclusion Criteria:

1. Demonstrates understanding of the study.
2. Aged 18 to 85 years.
3. Understands and is willing, able and likely to comply with all study procedures and restrictions.
4. Has good general health (in the opinion of the investigator or medically qualified designee).
5. A salivary flow-rate in the range of normal values (unstimulated whole saliva flow- Rate ≥ 0.2 g/minute (min); gum base stimulated whole saliva flow-Rate ≥ 0.8 g/min).
6. Currently wearing a removable mandibular partial denture with sufficient room in the posterior buccal flange area to accommodate two enamel specimens.
7. Have no current active caries or periodontal disease and all restorations in a good state of repair.
8. Willing and capable of brushing their natural teeth with the lower partial denture in place.

Exclusion Criteria:

1. Pregnant or breast feeding women.
2. Known or suspected intolerance or hypersensitivity to the study materials or their stated ingredients.
3. Currently taking antibiotics or have taken antibiotics in the two weeks prior to the screening visit.
4. Unable to measure product weights accurately using the assigned study scale as determined by the study staff as demonstrated.
5. Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.
6. Have received a professional fluoride treatment within 14 days of randomization to the first treatment.
7. Recent history (within the last year) of alcohol or other substance abuse.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one center in United States.
Pre-assignment Details: A total of 58 participants were screened, of which 45 participants were randomized and 42 completed the study.
Groups:
- Overall Study: This was a single-centre, randomized, blinded (examiner and laboratory analyst), placebo-controlled, 6-treatment, 4-period cross-over, incomplete block design, in situ caries study in healthy adults who wore a removable bilateral mandibular partial denture. Each participant received Test Product 1 (Dentifrice containing 0.425 % weight by weight (w/w) phytate, and 1150 parts per million [ppm] fluoride [F]), Test Product 2 (Dentifrice containing 0.85 % w/w phytate, and 1150 ppm fluoride), Test Product 3 (Dentifrice containing 0.85 % w/w phytate, 0.3% zinc chloride, 0.5% sodium citrate, and 1150 ppm fluoride), Reference Product 1 (0 ppm fluoride), Reference Product 2 (Dentrifrice containing 1150 ppm fluoride toothpaste and Reference Product 3 (Dentrifrice containing 0.3% zinc chloride , 0.5% sodium citrate, and 1150 ppm fluoride).
Period: Overall Study
Arm/Group | Overall Study
Started | 45
Received Test Product 1 | 29
Received Test Prodcut 2 | 28
Received Test Prodcut 3 | 28
Received Reference Product 1 | 29
Received Reference Product 2 | 28
Received Reference Product 3 | 28
Completed | 42
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants were included for baseline evaluation.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 24
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Surface Microhardness Recovery (SMHR) of Phyte (0% 0.425% and 0.85%) at 2 Weeks
Description: SMHR test was used to assess the changes in mineralization status of partially demineralized enamel specimens using a Wilson 2100 Hardness tester. SMH was determined by measuring the length of the indentations of enamel specimens. % SMHR was calculated from indentation length (micrometer [μm]) of sound enamel specimen at baseline (B), indentation length (μm) after in vitro demineralization(D), indentation length (μm) after intra-oral exposure (R): [D-R/D-B]*100.
Time Frame: Baseline upto 2 weeks
Population: Intent-to-treat (ITT) population, all participants who were randomized, received the study products at least once and provided at least one post-baseline assessment of efficacy. Number of participants who missed enamel specimens were: Test product 1- [1], Test product 2- [1], Reference Product 1- [1], and Reference Product 2- [1].
Measure: Mean (Standard Deviation); unit: % SMHR
Groups:
- Test Product 1: Participants brushed their natural teeth with a pre-wetted toothbrush and their assigned experimental dentifrice (containing 0.425 % phytate, 1150 ppm F) for one timed minute twice daily, ensuring the enamel specimens retained within their mouths were not directly brushed. Participants then rinsed their mouths with 15 milliliters (ml) of tap water for approximately 10 seconds (s).
- Test Product 2: Participants brushed their natural teeth with a pre-wetted toothbrush and their assigned experimental dentifrice (containing 0.85 % phytate, 1150 ppm F) for one timed minute twice daily, ensuring the enamel specimens retained within their mouths were not directly brushed. Participants then rinsed their mouths with 15ml of tap water for approximately 10s.
- Reference Product 1: Participants brushed their natural teeth with a pre-wetted toothbrush and their assigned reference dentifrice (containing 0 ppm fluoride) for one timed minute, ensuring the enamel specimens retained within their mouths were not directly brushed. Participants then rinsed their mouths with 15ml of tap water for approximately 10s.
- Reference Product 2: Participants brushed their natural teeth with a pre-wetted toothbrush and their assigned reference dentifrice (containing 1150ppm F) for one timed minute, ensuring the enamel specimens retained within their mouths were not directly brushed. Participants then rinsed their mouths with 15ml of tap water for approximately 10s.
Arm/Group | Test Product 1 | Test Product 2 | Reference Product 1 | Reference Product 2
Number analyzed (Participants) | 28 | 28 | 29 | 28
% SMHR | 25.53 (21.513) | 26.81 (18.059) | 7.41 (18.648) | 28.88 (21.046)
Statistical Analysis 1: Comparison: Test Product 1 vs Reference Product 2; Test type: Superiority or Other; p = 0.7603, ANCOVA — From ANCOVA: Participant (random), treatment & period (fixed), subject-level baseline SMH, period-level baseline SMH, subject-level pre-treatment acid challenge SMH and period-level pre-treatment acid challenge SMH (covariates); Mean Difference (Net) = -1.09, 95% CI 2-sided [-8.11 to 5.94] — Difference is first named treatment minus second named treatment such that positive difference favors the first named treatment
Statistical Analysis 2: Comparison: Test Product 2 vs Reference Product 2; Test type: Superiority or Other; p = 0.3555, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -3.30, 95% CI 2-sided [-10.34 to 3.74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test Product 1 vs Test Product 2; Test type: Superiority or Other; p = 0.5335, ANCOVA — ANCOVA: Participant (random), treatment & period (fixed), Participant-level baseline SMH, period-level baseline SMH, Participant-level pre-treatment acid challenge SMH and period-level pre-treatment acid challenge SMH (covariates); Mean Difference (Net) = 2.21, 95% CI 2-sided [-4.81 to 9.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Reference Product 1 vs Reference Product 2; Treatment comparison corresponding to qualifying criteria for the analysis; Test type: Superiority or Other; p < .0001, ANCOVA — From ANCOVA: Participant (random), treatment & period (fixed), Participant -level baseline SMH, period-level baseline SMH, Participant -level pre-treatment acidchallenge SMH and period-level pre-treatment acid challenge SMH (covariates); Mean Difference (Net) = 22.96, 95% CI 2-sided [16.02 to 29.90] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: % SMHR of 0.85% Phytate Compared to 0% Phytate, in Presence of 1150ppm Fluoride and 0.3% ZnCl2, 0.3% ZnCl2 Compared to 0% ZnCl2 in the Presence of 1150ppm Fluoride and 0.3% ZnCl2 Compared to 0% ZnCl2 in the Presence of 1150ppm Fluoride and 0.85% Phytate
Description: SMHR test was used to assess the changes in mineralization status of partially demineralized enamel specimens using a Wilson 2100 Hardness tester. SMH was determined by measuring the length of the indentations of enamel specimens. % SMHR was calculated from indentation length (μm) of sound enamel specimen at baseline (B), indentation length (μm) after in vitro demineralization(D), indentation length (μm) after intra-oral exposure (R): [D-R/D-B]*100.
Time Frame: Baseline upto 2 weeks
Population: ITT population, all participants who were randomized, received the study products at least once and provided at least one post-baseline assessment of efficacy. Number of participants who missed enamel specimens were: Test product 2- [1], Test product 3- [2], Reference Product 2- [1], and Reference Product 3- [1].
Measure: Mean (Standard Deviation); unit: % SMHR
Groups:
- Test Product 2: Participants brushed their natural teeth with a pre-wetted toothbrush and their assigned dentifrice (containing 0.85 % phytate, 1150 ppm F) for one timed minute twice daily, ensuring the enamel specimens retained within their mouths were not directly brushed. Participants then rinsed their mouths with 15ml of tap water for approximately 10s.
- Test Product 3: Participants brushed their natural teeth with a pre-wetted toothbrush and their assigned dentifrice (containing 0.85 % phytate, 1150 ppm F, 0.3% ZnCl2) for one timed minute, ensuring the enamel specimens retained within their mouths were not directly brushed. Participants then rinsed their mouths with 15ml of tap water for approximately 10s
- Reference Product 2: Participants brushed their natural teeth with a pre-wetted toothbrush and their assigned dentifrice (containing 1150ppm F) for one timed minute, ensuring the enamel specimens retained within their mouths were not directly brushed. Participants then rinsed their mouths with 15ml of tap water for approximately 10s.
- Reference Product 3: Participants brushed their natural teeth with a pre-wetted toothbrush and their assigned dentifrice (containing 1150ppm F, 0.3% ZnCl2) for one timed minute, ensuring the enamel specimens retained within their mouths were not directly brushed. Participants then rinsed their mouths with 15ml of tap water for approximately 10s.
Arm/Group | Test Product 2 | Test Product 3 | Reference Product 2 | Reference Product 3
Number analyzed (Participants) | 28 | 28 | 28 | 28
% SMHR | 26.81 (18.059) | 23.38 (20.177) | 28.88 (21.046) | 28.80 (20.830)

3. Secondary Outcome: Transverse Microradiography (TMR) Net Remineralization Change (ΔM) Value of Phytate (0% 0.452% and 0.85%) at 4 Weeks
Description: TMR was used to assess changes in the mineral status of partially demineralized enamel specimens. Lesions were analyzed at baseline and Integrated Mineral Loss (∆Z): (∆Z =(lesion depth x 87) - area under the curve [Area under the curve which relates volume % mineral at distances from the specimen surface with respect to section thickness]). After treatment a further section was taken from each lesion specimen for radiography assessment; ∆Z was calculated. The change which occurred in mineral content (∆M) of the lesions as a result of treatment was calculated by: ∆M= (baseline ∆Z - Post-treatment ∆Z).
Time Frame: Baseline upto 4 weeks
Population: ITT population, all participants who were randomized, received the study products at least once and provided at least one post-baseline assessment of efficacy. Number of participants who missed enamel specimens were: Test product 1- [1], Test product 2- [1], and Reference Product 2- [1].
Measure: Mean (Standard Deviation); unit: [%vol mineral x µm
Groups:
- Test Product 1: Participants brushed their natural teeth with a pre-wetted toothbrush and their assigned dentifrice (containing 0.425 % phytate, 1150 ppm F) for one timed minute, ensuring the enamel specimens retained within their mouths were not directly brushed. Participants then rinsed their mouths with 15ml of tap water for approximately 10s.
- Test Product 2: Participants brushed their natural teeth with a pre-wetted toothbrush and their assigned dentifrice (containing 0.85 % phytate, 1150 ppm F) for one timed minute, ensuring the enamel specimens retained within their mouths were not directly brushed. Participants then rinsed their mouths with 15ml of tap water for approximately 10s.
Arm/Group | Test Product 1 | Test Product 2 | Reference Product 1 | Reference Product 2
Number analyzed (Participants) | 28 | 27 | 29 | 28
[%vol mineral x µm | 3055.36 (1459.283) | 2772.96 (989.567) | 3849.83 (1978.088) | 2720.00 (1151.914)

4. Secondary Outcome: TMR Δm Value of 0.85% Phytate Compared to 0% Phytate, in the Presence of 1150ppm F and 0.3% ZnCl2, 0.3% ZnCl2 Compared to 0% ZnCl2 in the Presence of 1150ppm F and 0.3% ZnCl2 Compared to 0% ZnCl2 in the Presence of 1150ppm F and 0.85% Phytate
Description: as for outcome 3
Time Frame: Baseline upto 4 weeks
Population: ITT population, all participants who were randomized, received the study products at least once and provided at least one post-baseline assessment of efficacy. Number of participants who missed enamel specimens were: Test product 2 - [1], Test product 3 - [2], Reference Product 2 - [1] and Reference Product 3 [1].
Measure: Mean (Standard Deviation); unit: [%vol mineral x µm
Arm/Group | Test Product 2 | Test Product 3 | Reference Product 2 | Reference Product 3
Number analyzed (Participants) | 27 | 27 | 28 | 28
[%vol mineral x µm | 2772.96 (989.567) | 2733.33 (1051.738) | 2720.00 (1151.914) | 2421.25 (677.286)

5. Secondary Outcome: Enamel Fluoride Uptake (EFU) of All Study Formulation Variables
Description: The microdrill enamel biopsy technique was used to analyze the fluoride uptake by enamel. Each enamel specimen was mounted on the long axis of a drill attached to a microdrill and drilled to a depth of approximately 100 μm through the entire lesion (four cores per specimen). The enamel powder pooled from four drilling samples was then immediately analyzed for fluoride content using fluoride specific electrode and pH/ion meter. The amount of fluoride-uptake by enamel was calculated based on the amount of fluoride divided by the area of the enamel cores and expressed as μg/cm^2.
Time Frame: At Week 2
Population: ITT population, all participants who were randomized, received the study products at least once and provided at least one post-baseline assessment of efficacy. Number of participants who missed enamel specimens were: Test product1-[1], Test product2-[1], Test product3-[2], Reference Product1-[1], Reference Product2-[1] and Reference Product3-[1].
Measure: Mean (Standard Deviation); unit: μg/cm^2
Groups:
- Reference Product 1: Participants brushed their natural teeth with a pre-wetted toothbrush and their assigned dentifrice (containing 0 ppm fluoride) for one timed minute, ensuring the enamel specimens retained within their mouths were not directly brushed. Participants then rinsed their mouths with 15ml of tap water for approximately 10s.
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Reference Product 1 | Reference Product 2 | Reference Product 3
Number analyzed (Participants) | 28 | 28 | 28 | 29 | 28 | 28
μg/cm^2 | 5.35 (2.038) | 4.78 (2.655) | 5.02 (2.499) | 1.09 (0.397) | 5.87 (2.772) | 5.37 (2.384)

6. Secondary Outcome: Enamel Fluoride Uptake (EFU) of All Study Formulation Variables
Description: as for outcome 5
Time Frame: At Week 4
Population: ITT population, all participants who were randomized, received the study products at least once and provided at least one post-baseline assessment of efficacy. Number of participants who missed enamel specimens were: Test product1-[1], Test product2-[2], Test product3-[3], Reference Product1-[1], Reference Product2-[1] and Reference Product3-[1].
Measure: Mean (Standard Deviation); unit: μg/cm^2
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Reference Product 1 | Reference Product 2 | Reference Product 3
Number analyzed (Participants) | 28 | 27 | 27 | 29 | 28 | 28
μg/cm^2 | 12.28 (6.756) | 11.09 (6.336) | 14.16 (12.851) | 1.64 (0.974) | 15.29 (10.177) | 15.11 (10.180)

ADVERSE EVENTS:
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Reference Product 1 | Reference Product 2 | Reference Product 3
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/29 | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/28 | 0/28 | 0/29 | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 9/28 | 9/28 | 10/28 | 7/29 | 4/27 | 8/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product 1 (N=28) | Test Product 2 (N=28) | Test Product 3 (N=28) | Reference Product 1 (N=29) | Reference Product 2 (N=27) | Reference Product 3 (N=28)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product 1 (N=28) | Test Product 2 (N=28) | Test Product 3 (N=28) | Reference Product 1 (N=29) | Reference Product 2 (N=27) | Reference Product 3 (N=28)
GINGIVAL ERYTHEMA (Gastrointestinal disorders) | 2 | 3 | 2 | 1 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Gingival ulceration (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 2
Oral mucosal erythema (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gingival oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Leukoplakia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Device Failure (Product Issues) | 1 | 1 | 0 | 0 | 1 | 0
Injury Associated With Device (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Angular cheilitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.